CLINICAL TRIAL: NCT05119387
Title: Genetisk Studie av Amyotrofisk Lateral Sklerose (ALS)
Brief Title: Genetic Study of Amyotrophic Lateral Sclerosis in Norway
Acronym: GAIN
Status: Recruiting | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: ALS Norge (Unknown); Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018/1916
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Genetics; Amyotrophic Lateral Sclerosis; Neurology; Clinical genetics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals diagnosed with ALS: Individuals diagnosed with ALS that are being followed through the Norwegian health-care system. ALS patients ( probable or definite per El-Escorial criteria)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of genetic characteristics

SUMMARY:
The purpose of this study is to explore the genetic causes relevant for ALS development in Norway.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be asked to complete a small questionnaire regarding family history and have a blood sample withdrawn. Blood samples, questionnaires, clinical information and signed consent is send to Department of Medical Genetics, Telemark Hospital Trust were the genetic analysis is performed successively throughout the recruitment period. Patients can choose to have their genetic results returned in a diagnostic setting.

ELIGIBILITY:
Inclusion Criteria:

* Probable or definite ALS
* Eligible to consent

Exclusion Criteria:

- not competent to give consent

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with ALS that are being followed through the Norwegian health-care system.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Gene frequency | 2020-2030
  Number of patients with disease causing mutations in high penetrant ALS genes
New ALS genes | 2024-2030
  Identify new ALS genes in the Norwegian ALS population
Genetic risk factors | 2022-2030
  Identify genetic risk factors for ALS in Norway.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Høyer, Principal Investigator — Telemark Hospital Trust, Norway
Locations (17):
- Norway (17):
  - Haukeland University Hospital, Department of Neurology, Bergen
  - Nordland Hospital Trust, Department of Neurology, Bodø
  - Vestre Viken Hospital Trust, Department of Neurology, Drammen
  - Førde Hospital Trust, Department of Neurology, Førde
  - Østfold Hospital Trust, Department of Neurology, Grålum
  - Fonna Hospital Trust, Department of Neurology, Haugesund
  - Sørlandet Hospital Trust, Department of Neurology, Kristiansand
  - Innlandet Hospital Trust, Department of Neurology, Lillehammer
  - Akershus University Hospital, Department of Neurology, Lørenskog
  - Møre and Romsdal Hospital Trust, Department of Neurology, Molde
  - Nord-Trøndelag Hospital Trust, Department of Neurology, Namsos
  - Oslo University Hospital, Department of Neurology, Oslo
  - Telemark Hospital, Department of Neurology, Skien
  - Stavanger University Hospital, Department of Neurology, Stavanger
  - University hospital of North Norway, Department of Neurology, Tromsø
  - St. Olavs Hospital, Department of Neurology, Trondheim
  - Vestfold Hospital Trust, Department of Neurology, Tønsberg